CLINICAL TRIAL: NCT03706690
Title: A Phase III, Randomised,Double-Blind,Placebo-Controlled,Study of Durvalumab as Consolidation Therapy in Patients With Locally Advanced,Unresectable NSCLC, Who Have Not Progressed Following Definitive, Platinum-Based Chemoradiation Therapy
Brief Title: A Study of Durvalumab as Consolidation Therapy in Non-Small Cell Lung Cancer Patients
Acronym: PACIFIC-5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D933YC00001; 2018-002294-22 (EudraCT Number)
Record Dates: First submitted 2018-08-23; First posted 2018-10-16 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; Double-Blind; PD-L1; MEDI4736; Durvalumab; PFS; OS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor, excluding supply chain management personnel and unblinded monitors of site pharmacies, will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Durvalumab Therapy (Experimental): Durvalumab (PD-L1 monoclonal antibody)1500 mg every 4 weeks [q4w] intravenously [iv] until clinical progression/deterioration or confirmed radiological progression)
  Interventions: Drug: Durvalumab
- Placebo Therapy (Placebo Comparator): Placebo (matching placebo for infusion every 4 weeks iv until clinical progression/deterioration or confirmed radiological progression)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg every 4 weeks [q4w] intravenously [iv] until clinical progression/ deterioration or confirmed radiological progression.
  Other Names: MEDI4736
  Arms: Durvalumab Therapy
Other: Placebo — Matching placebo for infusion every 4 weeks iv until clinical progression/deterioration or confirmed radiological progression
  Arms: Placebo Therapy

SUMMARY:
This is a Phase III, randomised, double-blind, placebo-controlled, multicentre study assessing the efficacy and safety of durvalumab compared with placebo, as consolidation therapy in patients with locally advanced, unresectable, non-small cell lung cancer (Stage III), who have not progressed following definitive, platinum-based, chemoradiation therapy.

DETAILED DESCRIPTION:
Approximately 400 patients will be randomized in a 2:1 to receive treatment with durvalumab or placebo therapy. The primary objective of this study is to assess the efficacy of durvalumab treatment compared with placebo in terms of PFS.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Documented NSCLC and present with locally advanced, unresectable (Stage III) disease;
3. Receipt of concurrent or sequential chemoradiation therapy,
4. No progression following definitive, platinum-based, concurrent or sequential chemoradiation therapy
5. World Health Organization (WHO) PS of 0 or 1;
6. No prior exposure to any anti CTLA-4, anti-PD-1, anti-PD-L1, or anti PD L2 antibodies, excluding therapeutic anticancer vaccines
7. Adequate organ and marrow function required
8. Life expectancy of at least 12 weeks
9. Tumor PD-L1 status, with the Ventana SP263 PD-L1 IHC assay determined by a reference laboratory, must be known prior to randomization.
10. Tumour sample requirements are as follows: Provision of a tumour tissue sample (newly acquired sample <=3 months old is preferred, but an archived sample <=6 months old is acceptable) in a quantity sufficient to allow for analysis.

Exclusion Criteria:

1. History of allogeneic organ transplantation, or another primary malignancy, or active primary immunodeficiency.
2. Active or prior documented autoimmune or inflammatory disorders
3. Uncontrolled intercurrent illness that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent
4. Active infection including tuberculosis hepatitis B hepatitis C (HCV), or human immunodeficiency virus (positive human immunodeficiency virus [HIV] 1/2 antibodies).
5. Mixed small cell and NSCLC histology, sarcomatoid variant
6. Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 from the prior chemoradiation therapy.
7. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2027-02-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong General Hospital, Guangdong Lung Cancer Institute
Locations (69):
- China (22):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Linhai
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- Research Site, Hong Kong, Hong Kong
- India (6):
  - Research Site, Bangalore
  - Research Site, Bengaluru
  - Research Site, Karamsad
  - Research Site, Kolkata
  - Research Site, Nashik
  - Research Site, Vadodara
- Mexico (5):
  - Research Site, Culiacán
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, San Luis Potosí City
- Philippines (7):
  - Research Site, Bacolod
  - Research Site, Baguio City
  - Research Site, Cagayan de Oro
  - Research Site, Cebu
  - Research Site, Davao City
  - Research Site, Quezon City
  - Research Site, San Juan City
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Poznan
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- Russia (10):
  - Research Site, Kazan, Tatarstan
  - Research Site, Kirov
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saransk
  - Research Site, Volgograd
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Seoul
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Konya
  - Research Site, Malatya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Wu YL, Wu L, Bi N, Cil T, Ge H, Zhu Z, Wang CL, Zhang W, Lv D, Mingyan E, Sun J, Pan Y, Krzakowski M, Dikilitas M, Sendur MAN, Kim YC, Yang Y, Mao R, Zhang B, Wang L. PACIFIC-5: a phase III clinical trial of consolidation durvalumab in patients with unresectable stage III NSCLC and no progression after concurrent or sequential chemoradiotherapy. J Hematol Oncol. 2025 Dec 7;18(1):111. doi: 10.1186/s13045-025-01768-1. PMID 41354932
- See also: D933YC00001_CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933YC00001&attachmentIdentifier=5d25cd33-ab14-4e73-a7c7-6e0562df6739&fileName=D933YC00001_CSP_Redacted.pdf&versionIdentifier=
- See also: D933YC00001_CSR synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933YC00001&attachmentIdentifier=428778b4-8367-433e-944d-7fc6dfb71973&fileName=D933YC00001_CSR_synopsis_Redacted.pdf&versionIdentifier=
- See also: D933YC00001_SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933YC00001&attachmentIdentifier=04d4fd0e-ce5b-44cd-9255-db924c18e890&fileName=D933YC00001_SAP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III double-blind, placebo-controlled study was conducted at 82 investigational sites across 10 countries in participants with locally advanced, unresectable, non-small cell lung cancer (Stage III), who had not progressed following definitive, platinum-based, chemoradiation therapy (CRT).
Pre-assignment Details: The study consisted of a screening period (Day -84 to Day -1), randomization (Day 1), treatment period commencing on Day 1 and a survival follow-up period until protocol-specified discontinuation criteria were met. A total of 407 participants were randomized in a 2:1 ratio to receive either durvalumab or placebo in this study. Results are presented up to data cut-off (DCO) date of 23-Jun-2024.
Groups:
- Durvalumab: Participants received durvalumab 1500 milligram (mg) via intravenous (IV) infusion on Day 1 and every 4 weeks (Q4W) thereafter until confirmed radiological progression, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Placebo: Participants received placebo matched to durvalumab via IV infusion on Day 1 and Q4W thereafter until confirmed radiological progression, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
Period: Overall Study
Arm/Group | Durvalumab | Placebo
Started (Randomized) | 272 | 135
Participants Who Received Treatment | 271 | 134
Intent-to-treat (ITT) Set | 272 | 135
Modified Intent-to-treat (mITT) Set | 252 | 129
Completed | 0 | 0
Not Completed | 272 | 135
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Death | 143 | 75
Not completed — Ongoing at DCO | 121 | 52

BASELINE CHARACTERISTICS:
Population: The ITT set included all randomized participants.
Groups:
- Durvalumab: Participants received durvalumab 1500 mg via IV infusion on Day 1 and Q4W thereafter until confirmed radiological progression, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | Durvalumab | Placebo | Total
Number analyzed (Participants) | 272 | 135 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.33) | 61.9 (7.96) | 61.7 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 247 | 117 | 364
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 267 | 135 | 402
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 197 | 97 | 294
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 75 | 38 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) (Modified Intent-to-Treat [mITT] Set)
Description: The PFS per Response Evaluation Criteria in Solid Tumors 1.1. (RECIST 1.1) using blinded independent central review (BICR) assessments was defined as the time from the date of randomization until the date of objective disease progression (PD) or death (by any cause in the absence of progression) regardless of whether the participant withdrew from therapy or received another anti-cancer therapy prior to progression. The PD was defined as at least a 20% increase in the sum of diameters of target lesions (TLs) and an absolute increase of >=5 millimeters (mm), taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumor scans performed at screening, every 8 weeks ±1 week up to 48 weeks, and then every 12 weeks ±1 week thereafter until confirmed PD. Assessed up to the DCO date 23-Jun-2024 (a maximum of approximately 2035 days)
Population: The mITT set included all randomized participants who were without sensitizing epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) rearrangements.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 252 | 129
months | 14.0 [10.9 to 18.0] | 6.5 [5.4 to 13.8]
Statistical Analysis 1: Comparison: Durvalumab vs Placebo; The hazard ratio and confidence intervals (CIs) were calculated using a stratified Cox proportional hazards model, adjusting for the level of programmed death ligand 1 (PD-L1) expression (PD-L1 <1% versus [vs] PD-L1 >=1%) and prior therapy (concurrent [c]CRT vs sequential [s]CRT), with treatment as the only covariate and ties handled by Efron approach; Test type: Superiority; p = 0.038, Log Rank; Analysis performed using stratified log-rank test, adjusting for the level of PD-L1 expression and prior therapy (cCRT vs sCRT); Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.578 to 0.986]

2. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from the date of randomization until death due to any cause regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy. Median OS was calculated using the Kaplan-Meier technique.
Time Frame: Assessed up to the DCO date 23-Jun-2024 (a maximum of approximately 2035 days)
Population: Analysis was performed on the mITT and ITT set. The mITT set included all randomized participants who were without sensitizing EGFR mutations or ALK rearrangements. The ITT set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 272 | 135
months
  mITT set: number analyzed (Participants) | 252 | 129
  mITT set | 38.3 [28.9 to 42.8] | 32.5 [20.6 to 40.4]
  ITT set | 38.4 [29.0 to 42.9] | 32.5 [20.6 to 40.4]
Statistical Analysis 1: Comparison: Durvalumab vs Placebo; For mITT set. The hazard ratio and CIs were calculated using a stratified Cox proportional hazards model, adjusting for the level of PD-L1 expression (PD-L1 <1% vs PD-L1 >=1%) and prior therapy (cCRT vs sCRT), with treatment as the only covariate and ties handled by Efron approach; Test type: Superiority; p = 0.346, Log Rank; Analysis performed using stratified log-rank test, adjusting for level of PD-L1 expression and prior therapy (cCRT vs. sCRT); Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.656 to 1.166]
Statistical Analysis 2: Comparison: Durvalumab vs Placebo; For ITT set. The hazard ratio and CIs were calculated using a stratified Cox proportional hazards model, adjusting for the level of PD-L1 expression (PD-L1 <1% vs PD-L1 >=1%) and prior therapy (cCRT vs sCRT), with treatment as the only covariate and ties handled by Efron approach; Test type: Superiority; p = 0.346, Log Rank; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.663 to 1.162]

3. Secondary Outcome: Progression-Free Survival (PFS) (Intent-to-Treat [ITT] Set)
Description: The PFS per RECIST 1.1 using BICR assessments was defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdrew from therapy or received another anti-cancer therapy prior to progression. The PD was defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of >=5 mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 1
Population: The ITT set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 272 | 135
months | 14.1 [10.9 to 18.2] | 7.4 [5.5 to 13.8]
Statistical Analysis 1: Comparison: Durvalumab vs Placebo; The hazard ratio and CIs were calculated using a stratified Cox proportional hazards model, adjusting for the level of PD-L1 expression (PD-L1 <1% vs PD-L1>=1%) and prior therapy (cCRT vs sCRT), with treatment as the only covariate and ties handled by Efron approach; Test type: Superiority; p = 0.026, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.575 to 0.966]

4. Secondary Outcome: Percentage of Participants Alive at 24 Months (OS24)
Description: OS was defined as the time from the date of randomization until death due to any cause regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy. The OS24 was defined as the Kaplan-Meier estimate of OS at 24 months after randomization.
Time Frame: Month 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 272 | 135
percentage of participants
  mITT set: number analyzed (Participants) | 252 | 129
  mITT set | 60.7 [54.2 to 66.5] | 54.4 [45.2 to 62.7]
  ITT set | 60.8 [54.7 to 66.5] | 54.6 [45.6 to 62.8]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR per RECIST 1.1 using BICR was defined as the percentage of participants with at least 1 visit response of complete response (CR) or partial response (PR) based on all participants in the subset of the analysis population including only those participants with measurable disease at baseline per BICR. The CR was defined as disappearance of all TLs since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm. The PR was defined as at least a 30% decrease in the sum of the diameters of TLs, taking as reference the baseline sum of diameters as long as criteria for PD are not met.
Time Frame: as for outcome 1
Population: Analysis was performed on the mITT and ITT set. The mITT set included all randomized participants who were without sensitizing EGFR mutations or ALK rearrangements. The ITT set included all randomized participants. Only those participants with measurable disease at baseline per BICR are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 240 | 127
percentage of participants
  mITT set: number analyzed (Participants) | 221 | 121
  mITT set | 27.6 | 20.7
  ITT set | 27.1 | 19.7
Statistical Analysis 1: Comparison: Durvalumab vs Placebo; For mITT set. The comparison was performed using a logistic regression model, with treatment as a covariate and adjusting for the level of PD-L1 expression (PD-L1 <1% vs. PD-L1 >=1%) and prior therapy (cCRT vs. sCRT), with 95% CI calculated by profile likelihood; Test type: Superiority; p = 0.128, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.891 to 2.607]
Statistical Analysis 2: Comparison: Durvalumab vs Placebo; For ITT set. The comparison was performed using a logistic regression model, with treatment as a covariate and adjusting for the level of PD-L1 expression (PD-L1 <1% vs. PD-L1 >=1%) and prior therapy (cCRT vs. sCRT), with 95% CI calculated by profile likelihood; Test type: Superiority; p = 0.105, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.915 to 2.638]

6. Secondary Outcome: Duration of Response (DoR)
Description: The DoR per RECIST 1.1 using BICR was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of PD. PD was defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of >=5 mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters. The DoR was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 1
Population: Analysis was performed on the mITT and ITT set. The mITT set included all randomized participants who were without sensitizing EGFR mutations or ALK rearrangements. The ITT set included all randomized participants. Only responders (participants with objective response) are analyzed and reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 65 | 25
months
  mITT set: number analyzed (Participants) | 61 | 25
  mITT set | NA [16.6 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of participants with events at DCO date. | 37.6 [5.4 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at DCO date.
  ITT set | NA [20.7 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of participants with events at DCO date. | 37.6 [5.4 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at DCO date.

7. Secondary Outcome: Percentage of Participants Alive and Progression-Free at 12 and 18 Months (PFS12 and PFS18)
Description: The PFS per RECIST 1.1 using BICR assessments was defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdrew from therapy or received another anti-cancer therapy prior to progression. The PD was defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of >=5 mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters. The PFS12 and PFS18 were defined as the Kaplan-Meier estimate of PFS per RECIST 1.1 as assessed by the Investigator at 12 and 18 months, respectively and both were obtained using the algorithm for the RECIST 1.1 site Investigator tumor data.
Time Frame: Months 12 and 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 272 | 135
percentage of participants
  PFS12, mITT set: number analyzed (Participants) | 252 | 129
  PFS12, mITT set | 53.6 [47.0 to 59.7] | 42.7 [33.8 to 51.4]
  PFS18, mITT set: number analyzed (Participants) | 252 | 129
  PFS18, mITT set | 43.4 [36.9 to 49.7] | 34.1 [25.6 to 42.8]
  PFS12, ITT set | 54.2 [47.9 to 60.1] | 42.5 [33.8 to 51.0]
  PFS18, ITT set | 44.2 [37.9 to 50.3] | 33.4 [25.1 to 41.9]

8. Secondary Outcome: Time From Randomization to Second Progression (PFS2)
Description: PFS2 was defined as the time from the date of randomization to the earliest of the progression event subsequent to first subsequent therapy, or death. The date of the second progression was recorded by the Investigator and defined according to local standard clinical practice and could have involved any of objective radiological imaging, symptomatic progression, or death. Median time to PFS2 was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 272 | 135
months
  mITT set: number analyzed (Participants) | 252 | 129
  mITT set | 26.4 [22.1 to 36.0] | 19.5 [14.7 to 28.9]
  ITT set | 26.2 [22.0 to 34.8] | 19.5 [14.3 to 28.9]
Statistical Analysis 1: Comparison: Durvalumab vs Placebo; For mITT set. The hazard ratio and CIs were calculated using a stratified Cox proportional hazards model, adjusting for the level of PD-L1 expression (PD-L1 <1% vs. PD-L1 >=1%) and prior therapy (cCRT vs. sCRT), with treatment as the only covariate and ties handled by Efron approach; Test type: Superiority; p = 0.275, Log Rank; The analysis was performed using the stratified log-rank test, adjusting for the level of PD-L1 expression and prior therapy (cCRT vs. sCRT); Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.648 to 1.138]
Statistical Analysis 2: Comparison: Durvalumab vs Placebo; For ITT set. The hazard ratio and CIs were calculated using a stratified Cox proportional hazards model, adjusting for the level of PD-L1 expression (PD-L1 <1% vs. PD-L1 >=1%) and prior therapy (cCRT vs. sCRT), with treatment as the only covariate and ties handled by Efron approach; Test type: Superiority; p = 0.241, Log Rank; [statistical method as in outcome 8, analysis 1]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.648 to 1.122]

9. Secondary Outcome: Time to Death or Distant Metastases (TTDM)
Description: TTDM as per RECIST 1.1 using BICR was defined as the time from the date of randomization until the first date of distant metastasis or death in the absence of distant metastasis. Distant metastasis was defined as any new lesion that was outside of the radiation field according to RECIST 1.1. Median TTDM was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 272 | 135
months
  mITT set: number analyzed (Participants) | 252 | 129
  mITT set | 42.6 [33.2 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at DCO date. | NA [20.3 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of participants with events at DCO date.
  ITT set | 42.6 [33.2 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at DCO date. | NA [20.3 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of participants with events at DCO date.
Statistical Analysis 1: Comparison: Durvalumab vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.769, Log Rank; [statistical method as in outcome 8, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.726 to 1.578]
Statistical Analysis 2: Comparison: Durvalumab vs Placebo; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = 0.812, Log Rank; [statistical method as in outcome 8, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.726 to 1.539]

10. Secondary Outcome: Serum Concentration of Durvalumab
Description: Blood samples were collected to determine the concentration of durvalumab.
Time Frame: End of infusion on Cycle 1 Day 1, pre-infusion on Cycles 2 and 4 Day 1 and Month 3 follow-up (each cycle=28 days)
Population: The Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of durvalumab as per protocol for whom any post-dose data were available and who did not violate/deviate from protocol in ways that would significantly have affected the PK analyses. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Durvalumab
Number analyzed (Participants) | 249
nanogram/milliliter
  Cycle 1 Day 1 | 511415.541 (222137.0134)
  Cycle 2 Day 1: number analyzed (Participants) | 239
  Cycle 2 Day 1 | 93929.182 (86188.4708)
  Cycle 4 Day 1: number analyzed (Participants) | 205
  Cycle 4 Day 1 | 138752.016 (73792.7522)
  Month 3 follow-up: number analyzed (Participants) | 38
  Month 3 follow-up | 40303.562 (47725.6327)

11. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Durvalumab
Description: Blood samples were collected to determine the presence of ADAs and ADA-neutralizing antibodies (nAb) for durvalumab using validated assays. ADA prevalence was defined as the number of participants with positive ADA result at any time, baseline or post-baseline. ADA incidence was defined as either treatment-induced (post-baseline ADA positive only) or treatment-boosted ADA (baseline positive ADA titer that was boosted to >=4-fold during the study period). Treatment-induced ADA was defined as ADA positive only post-baseline and not detected at baseline. Persistently positive was defined as having at least 2 post-baseline ADA positive assessments with at least 16 weeks between the first and last positive assessment, or ADA positive at the last post-baseline assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive assessment without fulfilling the conditions for persistently positive.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2 and 4 (each cycle=28 days)
Population: ADA analysis set included all participants who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 255
Participants
  ADA positive at any visit (ADA prevalence) | 9
  Treatment-emergent ADA positive (ADA incidence) | 3
  ADA positive at both baseline and post-baseline | 1
  Treatment-induced ADA | 3
  ADA positive at baseline only | 5
  Treatment-boosted ADA | 0
  Persistently positive | 0
  Transiently positive | 4
  nAb positive | 2

12. Secondary Outcome: Change From Baseline in Patient-Reported Symptoms as Assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaires (EORTC QLQ) at Week 132
Description: Patient reported outcomes for 5 disease related symptoms was assessed using EORTC QLQ-Core 30 (C30) items questionnaire (fatigue, appetite loss) and EORTC QLQ-Lung Cancer module 13 (LC13) (dyspnoea, cough and pain in chest).An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items, functional scales, and global health status scale with higher scores on global health status/QoL and functioning scales representing better health status/function, but higher scores on symptom scales/items representing greater symptom severity. An improvement in symptoms were indicated by a negative change in score from baseline. A positive change in score from baseline indicated a deterioration of symptoms. A minimum clinically meaningful change was defined as change from baseline of >=10. Change from baseline in C30: global health status/QoL, physical functioning, fatigue, appetite loss and LC13: dyspnoea, cough and pain in chest are presented.
Time Frame: Baseline (Day 1) and Week 132
Population: Analysis was performed on the mITT and ITT set. The mITT set included all randomized participants who were without sensitizing EGFR mutations or ALK rearrangements. The ITT set included all randomized participants. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 63 | 22
units on a scale
  mITT set: EORTC QLQ-C30: Global health status/QoL: number analyzed (Participants) | 57 | 21
  mITT set: EORTC QLQ-C30: Global health status/QoL | 78.95 (13.918) | 74.21 (17.261)
  mITT set: EORTC QLQ-C30: Physical functioning: number analyzed (Participants) | 57 | 21
  mITT set: EORTC QLQ-C30: Physical functioning | 90.76 (10.216) | 92.38 (11.012)
  mITT set: EORTC QLQ-C30: Fatigue symptom: number analyzed (Participants) | 57 | 21
  mITT set: EORTC QLQ-C30: Fatigue symptom | 10.14 (13.814) | 13.76 (18.225)
  mITT set: EORTC QLQ-C30: Appetite loss symptom: number analyzed (Participants) | 57 | 21
  mITT set: EORTC QLQ-C30: Appetite loss symptom | 5.85 (12.791) | 3.17 (10.026)
  mITT set: EORTC QLQ-LC13: Dyspnoea symptom: number analyzed (Participants) | 57 | 21
  mITT set: EORTC QLQ-LC13: Dyspnoea symptom | 15.98 (14.998) | 11.11 (12.172)
  mITT set: EORTC QLQ-LC13: Cough symptom: number analyzed (Participants) | 57 | 21
  mITT set: EORTC QLQ-LC13: Cough symptom | 16.37 (21.009) | 22.22 (21.943)
  mITT set: EORTC QLQ-LC13: Pain in chest symptom: number analyzed (Participants) | 57 | 21
  mITT set: EORTC QLQ-LC13: Pain in chest symptom | 9.94 (16.625) | 6.35 (13.412)
  ITT set: EORTC QLQ-C30: Global health status/QoL | 78.70 (13.943) | 74.24 (16.846)
  ITT set: EORTC QLQ-C30: Physical functioning | 90.79 (10.120) | 92.73 (10.869)
  ITT set: EORTC QLQ-C30: Fatigue symptom | 10.93 (14.866) | 13.13 (18.026)
  ITT set: EORTC QLQ-C30: Appetite loss symptom | 5.29 (12.279) | 3.03 (9.808)
  ITT set: EORTC QLQ-LC13: Dyspnoea symptom | 15.17 (14.974) | 10.61 (12.112)
  ITT set: EORTC QLQ-LC13: Cough symptom | 15.87 (21.467) | 21.21 (21.932)
  ITT set: EORTC QLQ-LC13: Pain in chest symptom | 10.05 (17.592) | 7.58 (14.298)

13. Secondary Outcome: Number of Participants With Positive Programmed Death Ligand 1 (PD-L1) Status Based on Overall Survival, Progression-Free Survival and Objective Response Rate
Description: Blood samples will be collected for clinical biomarker testing and a tumor specimen will be collected as per tumor specimen collection requirements. The specimen will be evaluated by immunohistochemistry to determine the expression of tumor specific antigens and immune markers. The PD-L1 is a biomarker and data for number of participants with its positive status will be presented.
Time Frame: Up to 9 years
Reporting Status: Not Posted, anticipated posting 2027-03

ADVERSE EVENTS:
Time Frame: From time of signature of informed consent up to the DCO date 23-Jun-2024 (a maximum of approximately 2035 days)
Description: The Safety analysis set included all participants who received at least 1 dose of study treatment. All-cause mortality was determined for all randomized participants.
Arm/Group | Durvalumab | Placebo
All-Cause Mortality (participants affected / at risk) | 143/272 | 75/135
Serious Adverse Events (participants affected / at risk) | 104/271 | 45/134
Other Adverse Events (participants affected / at risk) | 223/271 | 94/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=271) | Placebo (N=134)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal-pulmonary fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 2 (4)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 21 (23) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 6 (7) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 14 (14) | 12 (12)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Myocardial injury (Cardiac disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 4 (4) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Victim of homicide (Social circumstances) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=271) | Placebo (N=134)
Fatigue (General disorders) | 18 (20) | 4 (4)
Pyrexia (General disorders) | 14 (19) | 5 (7)
Hepatic function abnormal (Hepatobiliary disorders) | 14 (15) | 2 (2)
COVID-19 (Infections and infestations) | 30 (31) | 13 (13)
Herpes zoster (Infections and infestations) | 7 (8) | 9 (9)
Pneumonia (Infections and infestations) | 35 (37) | 11 (11)
Anaemia (Blood and lymphatic system disorders) | 41 (57) | 20 (27)
Upper respiratory tract infection (Infections and infestations) | 30 (40) | 15 (20)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 52 (53) | 27 (27)
Alanine aminotransferase increased (Investigations) | 27 (43) | 6 (8)
Amylase increased (Investigations) | 22 (44) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 25 (48) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 16 (17) | 11 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (28) | 5 (7)
Hyperuricaemia (Metabolism and nutrition disorders) | 16 (32) | 4 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (9) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (23) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (20) | 6 (6)
Insomnia (Psychiatric disorders) | 14 (15) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (37) | 15 (17)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (11)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 6 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (22) | 6 (6)
Hyperthyroidism (Endocrine disorders) | 33 (41) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 21 (27) | 9 (11)
Hypothyroidism (Endocrine disorders) | 51 (67) | 10 (13)
Constipation (Gastrointestinal disorders) | 16 (17) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 14 (16) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT03706690/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03706690/SAP_001.pdf